

## STUDY PROTOCOL

(June 30th 2019)

# The Role of Beta-1,3/1,6-D-Glucan from Mycelium Extract of Indonesian *Ganoderma Lucidum* on Ulcerative Colitis: A Double-Blind Randomized Controlled Trial

PRINCIPAL INVESTIGATOR: Prof. dr. Marcellus Simadibrata, PhD., SpPD-KGEH

CO-INVESTIGATOR : Prof. Dr. dr. Murdani Abdullah, SpPD-KGEH

dr. Rabbinu Rangga Pribadi, SpPD

**Faculty of Medicine** 

**Universitas Indonesia** 

(FMUI)

#### Title

The Role of Beta-1,3/1,6-D-Glucan from Mycelium Extract of Indonesian Ganoderma Lucidum on Ulcerative Colitis: A Double-Blind Randomized Controlled Trial

## Background

Inflammatory bowel disease (IBD) is an autoimmune disorder there is marked by chronic inflammation in gastrointestinal system.<sup>1</sup> IBD is classified to two types, ulcerative colitis (UC) and Crohn's disease (CD). These are based on difference pathology and clinical manifestation. The common symptom of IBD is chronic diarrhoea with or without blood, abdominal cramp and weight loss.<sup>2,3</sup> IBD has high incidence and prevalence in Europe and America. Incidence of UC and CD in Europe are 24.3 and 29.3 by 100,000 respectively.<sup>4</sup> On the last few decades, there was an increasing incidence and prevalence IBD on Asia and other developing countries.<sup>5</sup> In Indonesia, incidence of UC and CD are 0.55 and 0.33 by 100.0000 respectively.<sup>6</sup> Trends in epidemiology of IBD was related to westernized lifestyle, urbanization, and hygiene as a part of socioeconomic development in developing countries.<sup>7</sup>

Nowadays, IBD treatment focus to prevent complication, maintain remission phase and improve quality of life. Drugs that are widely used for improving symptoms of IBD are anti-inflammatory drugs (5-aminosalicylic acid), immunomodulator (azathioprine, mercaptopurine, methotrexate), and biologic agent. These drugs work by increasing Th2-mediated response that cause a decrease in inflammation mediated by Th1.<sup>8</sup> Long term use of these drugs will cause different side effects. Side effects from immunomodulator are myelosuppression, hepatitis and increase risk of malignancy. Use of anti TNF-α will cause lupus like syndrome and malignancy.<sup>9</sup> Therefore, we need alternative treatment of IBD that effective but minimal side effects.

Ganoderma lucidum is a species from Ganodermataceae family that has Beta-1,3/1,6-D-Glucan as one of active compound from isolated mycelium extract Ganoderma lucidum. This compound has biologic effect as immunomodulator and has been used to prevent and treat diseases such as gastric ulcer, arthritis, atherosclerosis, asthma, diabetes, cancer and other diseases related to immune disorders. A study on patient with CD showed that Ganoderma lucidum decrease TNF- $\alpha$ , IFN- $\gamma$ , IL-17A from inflammation of intestinal mucosa. On the other hand, there is no study about the role of Beta-1,3/1,6-D-Glucan Ganoderma lucidum in UC.

## **Objective**

## General objective

To know the role of Beta-1,3/1,6-D-Glucan from mycelium extract of Ganoderma lucidum administration in ulcerative colitis

## Specific objectives

- 1. To know the quality of life from patient with ulcerative colitis after Beta-1,3/1,6-D-Glucan mycelium extract of Ganoderma lucidum administration
- 2. To know the level of inflammatory marker from patient with ulcerative colitis after Beta-1,3/1,6-D-Glucan mycelium extract of Ganoderma lucidum administration
- 3. To know the Mayo score from patient with ulcerative colitis after Beta-1,3/1,6-D-Glucan mycelium extract of Ganoderma lucidum administration

#### Methods

## Study Design

This research is a double blind, randomized clinical trial method. Analysis will be conducted pre and post administration: control (placebo) and intervention (polysaccharide peptide Ganoderma lucidum) 3 times daily for 90 days.

#### **Location and Time**

This research will be conducted on Indonesia from August 2019 to December 2020

#### Population and Subject

#### **Population**

The population of this research is patients diagnosed with ulcerative colitis in Indonesia

#### Subjects Criteria

- Inclusion criteria
  - 1. Subjects aged  $\geq$  18 years old
  - 2. Ulcerative colitis patients who are treated by 5-ASA 3x500 mg
  - 3. Agreed to participate

#### - Exclusion criteria

1. Allergic with Ganoderma lucidum

- 2. Ulcerative colitis patients who are treated by corticosteroid, immunosuppressive agent, biologic agent
- 3. Could not be randomised and participate in this study by clinical judgement

## Drop Out Criteria

Drop out subjects are subjects who have signed the informed consent but decide to withdraw before research is completed

## **Estimated Sample Size**

Minimum sample size is determined using the following equation for proportion equation.

N1 = N2 = 
$$\frac{(Z_{\alpha}\sqrt{2PQ} + Z_{\beta}\sqrt{P_1Q_1 + P_2Q_2})^2}{(P_1 - P_2)^2}$$

Description:

$$Z\alpha = 1.96 \qquad Z\beta = 0.84$$
 
$$P_1 \text{-} P_2 = 0.2 \qquad P_1 = 0.554^{12}$$

N1 = N2 = 92.25, thus with predicted drop out 10% the minimal sample for each group is 102 subjects

# Randomization

Randomization is generated by computer and subjects will be given code and divided into two groups (control and intervention). Researcher and subjects are blinded to treatment.

#### <u>Variables</u>

#### **Independent Variables**

- 1. Intervention: administration of capsule contain Beta-1,3/1,6-D-Glucan as active form of polysaccharide peptide from mycelium extract *Ganoderma lucidum* 3 times daily
- 2. Control (placebo): administration of empty capsule 3 times daily

## Dependent Variables

- 1. Quality of life; assessed by Indonesian validated SF-36 questionnaire
- 2. Erythrocyte Sedimentation Rate (ESR), C-Reactive Protein (CRP), Tumor Necrosis Factor Alpha (TNF-α) and Interleukin 6 (IL-6) from blood samples

- 3. Fecal calprotectin from stool examination
- 4. Mayo Score from colonoscopy
- 5. Biopsy

## Procedure

1. Eligibility assessment

The subjects will be assessed for eligibility using inclusion and exclusion criteria.

- 2. Subjects sign the informed consent form
- 3. Randomization
- 4. Pre-administration

Before administration of polysaccharide peptide or placebo based on randomization, subjects will be analysed for his/her quality of life by SF 36 questionnaire, ESR, CRP, TNF- $\alpha$ , IL-6, fecal calprotectin, colonoscopy (Mayo Score) and biopsy.

5. Administration (90 days)

Subjects will be given *Ganoderma lucidum* and placebo that will be taken three times daily for 90 days. The drugs are given monthly to the subjects.

6. Compliance monitoring

Compliance monitoring of administration is conducted by the investigators coordinating with his/her family and checked monthly when the patients came to take the capsule for the next month

7. Post administration

After 90 days the subjects will be analysed for his/her quality of life by SF 36 questionnaire, ESR, CRP, TNF-α, IL-6, fecal calprotectin, colonoscopy (Mayo Score) and biopsy.

- 8. Data analysis
  - a. Normality analysis using Kolmogorov-Smirnov (Normally distributed if p>0.05)
  - Bivariate analysis by comparing numeric data between two groups: if data is normality distributed using T-test, if not using Mann-Whitney test (significant if p<0.05)</li>
  - c. Bivariate analysis by comparing categorical data between two groups: if data is normality distributed using T-test, if not using Mann-Whitney test (significant if p<0.05)

- d. Bivariate analysis by comparing numeric data between preadministration and postadministration: if data is normality distributed using paired T-test, if not using Wilcoxon test (significant if p<0.05)</li>
- e. Bivariate analysis by comparing categorical data between preadministration and postadministration: if data is normality distributed using Mc Nemar test, if not using Wilcoxon test (significant if p<0.05)

## Study flow chart



## Ethical committee approval

Approval from the Ethical Committee at the Faculty of Medicine Universitas Indonesia must be obtained before starting the trial.

#### References

- 1. Fakhoury M, Negrulj R, Mooranian A, Al-salami H. Inflammatory bowel disease: clinical aspects and treatments. *J Inflamm Res*. 2014;7:113-120.
- 2. Ye Y, Pang Z, Chen W, Ju S, Zhou C. The epidemiology and risk factors of inflammatory bowel disease. *Int J Clin Exp Med*. 2015;8(12):22529-22542.
- 3. Zhang H, An C, Jennifer AH, Nolan K. Bioactive dietary peptides and amino acids in inflammatory bowel disease. 2014.
- 4. Molodecky NA, Soon IS, Rabi DM, et al. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. *Gastroenterology*. 2012;142(1):46-54.e42.
- 5. Ng WK, Wong SH, Ng SC. Changing epidemiological trends of inflammatory bowel disease in Asia. *Intest Res.* 2016;14(2):111-119.
- 6. Ng SC, Tang W, Ching JY, et al. Incidence and phenotype of inflammatory bowel disease based on results from the Asia-Pacific Crohn's and colitis epidemiology study. *Gastroenterology*. 2013;145(1):158-165.
- 7. Ng SC. Epidemiology of Inflammatory Bowel Disease: Focus on Asia. *Best Pract Res Clin Gastroenterol*. 2014.
- 8. Burger D, Travis S. Conventional medical management of inflammatory bowel disease. *Gastroenterology*. 2011;140(6):1827-1837.
- 9. Liu C, Dunkin D, Lai J, Song Y, Benkov K, Li X. Anti-inflammatory Effects of Ganoderma Lucidum Triterpenoid in Human Crohn's Disease Associated with Down-Regulation of NF-KB Signaling. *Inflamm Bowel Dis.* 2016;21(8):1918-1925.
- 10. Jin M, Zhu Y, Shao D, et al. Effects of polysaccharide from mycelia of Ganoderma lucidum on intestinal barrier functions of rats. *Int J Biol Macromol*. 2017;94:1-9.
- 11. Wang C, Shi S, Chen Q, et al. Antitumor and Immunomodulatory Activities of Ganoderma lucidum Polysaccharides in Glioma-Bearing Rats. *Integr Cancer Ther*. 2018;(29).
- 12. Damiao AOMC, Azevedo MFC, Carlos AS, Wada MY, Silva TVM, Feitosa FC. Conventional therapy for moderate to severe inflammatory bowel disease: A systematic literature review. *World J Gastroenterol*. 2019;25(9):1142-1157